CLINICAL TRIAL: NCT01789840
Title: Prospective, Controlled Investigation of Prostate Artery Embolization With Embosphere Microspheres Compared to Transurethral Resection of the Prostate for the Treatment of Symptomatic Benign Prostatic Hyperplasia
Brief Title: Prostate Artery Embolization With Embosphere Microspheres Compared to TURP for Benign Prostatic Hyperplasia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: 510(K) Approval Gained for Product
Sponsor: Merit Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BPH-P3-12-01; 2012-003446-33 (EudraCT Number)
Record Dates: First submitted 2013-02-08; First posted 2013-02-12 (Estimated); Results first posted 2021-11-11 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-10

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: BPH; Prostate; Prostatic Hyperplasia; enlarged prostate; LUTS; urinary retention
MeSH Terms: conditions — Prostatic Hyperplasia; Urinary Retention | interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prostate artery embolization (PAE) (Experimental): Prostate artery embolization using Embosphere Microspheres
  Interventions: Device: Embosphere Microspheres
- Transurethral resection of the prostate (TURP) (Active Comparator): Transurethral Resection of the Prostate (TURP)
  Interventions: Procedure: TURP

INTERVENTIONS:
Device: Embosphere Microspheres
  Arms: Prostate artery embolization (PAE)
Procedure: TURP
  Other Names: TURP - Transurethral resection of the prostate
  Arms: Transurethral resection of the prostate (TURP)

SUMMARY:
The purpose of this study is to evaluate improvement of symptoms from benign prostatic hyperplasia (BPH) as assessed by the International Prostate Symptom Score (IPSS) for prostatic artery embolization (PAE) using Embosphere Microspheres compared to conventional transurethral resection of the prostate (TURP).

DETAILED DESCRIPTION:
The study will consist of a screening period in which patient eligibility will be determined and baseline assessments performed. Once eligibility is confirmed, patients will be enrolled within 4 weeks of baseline imaging to receive either TURP or PAE with Embosphere Microspheres. After treatment, patients will return for follow-up visits at Months 1, 3, 6, and 12. At each of these visits patients will complete IPSS and IIEF questionnaires and have a physical exam, laboratory assessments (including PSA), a DRE, and a transrectal ultrasound of the prostate. At each visit patients will have a cystoscopy and proctoscopy if medically indicated. Cystoscopy is necessary in all cases of hematuria (injury associated with bleeding). Proctoscopy is necessary in all cases of bleeding per the rectum. An MRI of the prostate will be conducted at the 3 and 12 month visits. Uroflowmetry testing will be performed at the 1 and 12 month visits, and at other visits if medically indicated. MRIs will be assessed by blinded Central Reviewers.

The primary endpoint will be improvement of symptoms from BPH evaluated using the IPSS at 12 months post treatment. Patients will continue to be followed annually for up to 4 additional years. At a minimum, patients will be requested to complete the IPSS and International Index of Erectile Dysfunction (IIEF) questionnaires by telephone, email or mail once per year during this long term follow up period. Patients who are willing to return to the clinic will have a physical exam, MRI of the prostate, digital rectal exam (DRE), transrectal ultrasound of the prostate, PSA, and uroflowmetry testing performed each year. Treatments for LUTS due to BPH after the study treatment and 12 month follow up are complete will be documented during the long term follow up period to the extent possible. This long term follow up data will be summarized and submitted separately from the data for the initial 12 months of this study.

Safety will be evaluated throughout the initial 12 months of the study by assessing adverse events, as well as changes in laboratory values, and findings on physical examination. Concomitant medication usage will be assessed. A follow up ECG will be performed at the 12 month visit.

Patient recruitment is anticipated to take approximately 2 years. Duration of each patient's participation is expected to be 5 years, including a 4 year long term follow up period. The total duration of the study will be approximately 7 years, including long term follow up.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is age 50 to 79, inclusive
2. Patient has signed informed consent
3. Patient has had lower urinary tract symptoms (LUTS) secondary to BPH for at least 6 months prior to study treatment
4. Patient has a baseline IPSS Score > 13 at baseline
5. Patient has a prostate size of at least 50 grams and not more than 90 grams, measured by MRI
6. Patient has BPH symptoms refractory to medical treatment or for whom medication is contraindicated, not tolerated or refused
7. Patient must be a candidate for TURP
8. Patient must meet one of the following criteria:

   * Baseline Prostate Specific Antigen (PSA) <2.5 ng/mL (no prostate biopsy required)
   * Baseline PSA >2.5 ng/mL and ≤10 ng/mL AND free PSA > 25% of total PSA (no prostate biopsy required)
   * Baseline PSA >2.5 ng/mL and ≤10 ng/mL AND free PSA < 25% of total PSA AND a negative prostate biopsy result (minimum 12 core biopsy)
   * Baseline PSA >10 ng/mL AND a negative prostate biopsy (minimum 12 core biopsy)

Exclusion Criteria:

1. Active urinary tract infection
2. Biopsy proven prostate or bladder cancer, or any cancer other than basal or squamous cell skin cancer

   * The following patients must undergo prostate biopsy with a minimum of 12 cores and have a negative histopathology report to be enrolled in the study:

     * Patients with digital rectal examination (DRE) findings suspicious for prostate cancer
     * Patients with baseline PSA levels > 10 ng/mL
     * Patients with baseline PSA levels >2.5 ng/mL and < 10ng/mL AND free PSA < 25% of total PSA
   * Patients with cystoscopy findings suspicious for bladder cancer must undergo biopsy and have a negative histopathology report to be enrolled in the study
3. Bladder atonia, neurogenic bladder disorder or other neurological disorder that is impacting bladder function (eg multiple sclerosis, Parkinson's disease, spinal cord injuries, etc)
4. Urethral stricture, bladder neck contracture, sphincter abnormalities, urinary obstruction due to causes other than BPH, or other potentially confounding bladder or urethral disease or condition
5. Patient has taken beta blockers, antihistamines, anticonvulsants, or antispasmodics within 1 week of study treatment AND has not been on the same drug dosage for 6 months with a stable voiding pattern

   • Dosage of these medications should not change during study participation unless medically necessary
6. Patient has taken antidepressants, anticholinergics, androgens or gonadotropin-releasing hormonal analogues within 2 months of study treatment AND has not been on the same drug dosage for at least 3 months with a stable voiding pattern
7. Patient has taken 5-alpha reductase inhibitors or alpha blockers within 1 month of study treatment AND has not been on the same drug dosage for at least 3 months with a stable voiding pattern
8. Previous non-medical BPH treatment, including surgery, TURP, needle ablation, microwave or laser therapy, balloon dilation, stent implantation, or any other invasive treatment to the prostate
9. Any known condition that limits catheter-based intervention or is a contraindication to embolization, such as intolerance to a vessel occlusion procedure or severe atherosclerosis.
10. Patient is unable to stop taking anticoagulant, nonsteroidal antiinflammatory drug (NSAID) or anti-platelet therapy for 7 days prior to study treatment
11. Unable to have MRI imaging (eg metal implant including pacemaker, replacement joint, etc)
12. Patient has an asymmetric prostate, with > 20% difference in size between lobes
13. Cardiac condition including congestive heart failure or arrhythmia, uncontrolled diabetes mellitus, significant respiratory disease or known immunosuppression which required hospitalization within the previous 6 months
14. Baseline serum creatinine level > 1.8 mg/dl
15. Known upper tract renal disease
16. Cystolithiasis or chronic hematuria within 3 months prior to study treatment
17. Active prostatitis
18. Previous rectal surgery other than hemorrhoidectomy, or history of rectal disease
19. History of pelvic irradiation or radical pelvic surgery
20. Patient is interested in future fertility
21. Coagulation disturbances not normalized by medical treatment
22. Acute urinary retention requiring an indwelling catheter
23. Known major iliac arterial occlusive disease
24. Allergy to iodinated contrast agents
25. Hypersensitivity to gelatin products

Ages: 50 Years to 79 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Francisco, Cesar Carnevale, PhD, Principal Investigator — University of Sao Paolo, Brazil
Locations (10):
- United States (10):
  - Long Beach VA, Long Beach, California
  - VA Greater Los Angeles Healthcare System, Los Angeles, California
  - Stanford University Medical Center, Stanford, California
  - Georgetown University Hospital, Washington D.C., District of Columbia
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Miami VA Healthcare System, Miami, Florida
  - University of Miami Hospital, Miami, Florida
  - Tampa General Hospital, Tampa, Florida
  - Johns Hopkins Medical Center, Baltimore, Maryland
  - Mount Sinai Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Prostate Artery Emoblization (PAE): Prostate artery embolization using Embosphere Microspheres
  Embosphere Microspheres
- Transurethral Resection of the Prostate (TURP): Transurethral Resection of the Prostate (TURP)
  TURP
Period: Overall Study
Arm/Group | Prostate Artery Emoblization (PAE) | Transurethral Resection of the Prostate (TURP)
Started | 52 | 7
Completed | 52 | 6
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Population: Clinical trial results analyzed when study was ongoing and at time of De Novo submission. Trial was terminated when De Novo clearance was obtained. No further analysis was performed and IDE was terminated. Baseline characteristics are presented for all enrolled subjects at time of study termination.
Groups:
- Total: Total of all reporting groups
Arm/Group | Prostate Artery Emoblization (PAE) | Transurethral Resection of the Prostate (TURP) | Total
Number analyzed (Participants) | 52 | 7 | 59
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.2 (6.73) | 62.9 (76.74) | 64.9 (6.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 52 | 7 | 59
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 2 | 14
  Not Hispanic or Latino | 40 | 5 | 45
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 1 | 0 | 1
  White | 47 | 7 | 54
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
International Prostate Symptom Score (IPSS) [Mean (Standard Deviation); unit: units on a scale] — The International Prostate Symptom Score (I-PSS) is based on the answers to seven questions concerning urinary symptoms and one question concerning quality of life. Each question concerning urinary symptoms allows the patient to choose one out of six answers indicating increasing severity of the particular symptom. The answers are assigned points from 0 to 5. The total score can therefore range from 0 to 35 (asymptomatic to very symptomatic). Mild is generally less than or equal to 7, moderate is 8-19 and severe is 20-35.
  units on a scale | 22.2 (5.25) | 24.6 (5.59) | 22.4 (5.30)
Peak Urine Flow Rate (Qmax reported as mL/s) [Mean (Standard Deviation); unit: mL/s] — Population: Deviation recorded for Qmax not performed on 1 subject at baseline
  mL/s
    number analyzed (Participants) | 51 | 7 | 58
    (all) | 6.6 (4.03) | 8.1 (3.98) | 6.7 (4.02)
Post Void Residual (PVR) [Mean (Standard Deviation); unit: mL] | 170.6 (156.27) | 112.0 (165.35) | 163.7 (157.06)
Detrusor Pressure (Pdet) (mmH2O) [Mean (Standard Deviation); unit: mmH2O] — Population: Protocol deviations recorded for Pdet not captured on 2 patients.
  mmH2O
    number analyzed (Participants) | 50 | 7 | 57
    (all) | 88.3 (71.25) | 80.9 (38.69) | 87.4 (67.99)
International Index of Erectile Function (IIEF) - Total [Mean (Standard Deviation); unit: units on a scale] — Q1-5 refer to erectile function. Q6-8 refer to satisfaction with intercourse. Q9-10 refer to orgasmic function. Q11-12 ask about sexual desire. Q13-14 refer to overall sexual satisfaction. Q15 refers to erectile function. Q1-5 &15 range from 0-5 (max score 30). Q 9-10 range from 0-5 (max score 10). Q11-12 range from 1-5 (max score 10). Q6-8 range from 0-5 (max score 15). Q13-14 range from 1-5 (max score 10).
  Erectile function score (Q1-5 & 15): 1-10=severe, 11-16=moderate, 17-21=mild-moderate, 22-25=mild, 26-30=no dysfunction. Total IIEF out of 75 pts, higher scores = less dysfunction
  units on a scale
    Total IIEF | 29.5 (20.71) | 48.6 (24.73) | 31.8 (21.89)
    Erectile function sub-score | 11.7 (9.82) | 20.1 (10.99) | 12.7 (10.25)
    Orgasmic function sub-score | 4.2 (3.76) | 5.7 (4.11) | 4.4 (3.81)
    Sexual desire sub-score | 5.1 (2.47) | 7.4 (2.70) | 5.4 (2.59)
    Intercourse satisfaction sub-score | 4.1 (4.63) | 8.0 (6.08) | 4.5 (4.93)
    Overall satisfaction sub-score | 4.5 (2.79) | 7.3 (3.30) | 4.8 (2.97)
Prostate volume (g) [Mean (Standard Deviation); unit: g] | 66.4 (11.8) | 65.9 (14.71) | 66.4 (12.04)
Prostate Specific Antigen (PSA) (ng/mL) [Mean (Standard Deviation); unit: ng/mL] | 3.9 (2.71) | 5.5 (6.71) | 4.1 (3.37)
Free Prostate Specific Antigen (PSA) [Mean (Standard Deviation); unit: percentage of Free PSA] — Population: Free PSA was not collected at baseline on all subjects due to protocol deviation
  percentage of Free PSA
    number analyzed (Participants) | 45 | 2 | 47
    (all) | 22.5 (8.99) | 21.8 (9.65) | 22.4 (8.91)

OUTCOME MEASURES:

1. Primary Outcome: International Prostate Symptom Score (IPSS) - Total Score at 12 Months
Description: The International Prostate Symptom Score (I-PSS) is based on the answers to seven questions concerning urinary symptoms and one question concerning quality of life. Each question concerning urinary symptoms allows the patient to choose one out of six answers indicating increasing severity of the particular symptom. The answers are assigned points from 0 to 5. The total score can therefore range from 0 to 35 (asymptomatic to very symptomatic). Mild is generally less than or equal to 7, moderate is 8-19 and severe is 20-35. Total score was measured at 12 months.
Time Frame: 12 months
Population: Merit Medical received 513(f)(2) (de novo) classification from the FDA expanding the indication for Embosphere Microspheres to include prostatic artery embolization (PAE) for symptomatic benign prostatic hyperplasia (BPH) in 2017. An IDE supplement was submitted for this study proposing the termination of study follow-up visits. The FDA granted approval of termination on 03 Nov 2017. Early termination resulted in small numbers analyzed, incomplete enrollment and follow-up of study subjects.
Measure: Mean (Standard Deviation); unit: total score on a scale
Arm/Group | Prostate Artery Emoblization (PAE) | Transurethral Resection of the Prostate (TURP)
Number analyzed (Participants) | 10 | 4
total score on a scale | 10.7 (8.8) | 4.3 (5.9)

2. Secondary Outcome: Duration of Hospitalization Post Procedure
Description: The duration of hospitalization associated with the procedure will be calculated in hours. T
Time Frame: 1 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Prostate Artery Emoblization (PAE) | Transurethral Resection of the Prostate (TURP)
Number analyzed (Participants) | 28 | 6
hours | 23.1 (9.4) | 32.2 (10.2)

3. Secondary Outcome: Duration of Post Procedure Catheterization
Description: The duration of post procedure catheterization will be calculated in hours.
Time Frame: 1 month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Prostate Artery Emoblization (PAE) | Transurethral Resection of the Prostate (TURP)
Number analyzed (Participants) | 27 | 6
hours | 24.2 (44.2) | 24.2 (12.9)

4. Secondary Outcome: Number of Adverse Events Per Patient
Description: Adverse events during the study were predominantly mild. There are over 4 times as many PAE patients as TURP, so the overall incidence rate of events is proportional to the size of the cohort represented. The most common events among patients who underwent embolization were transient dysuria, bladder spasm, hematuria, hematospermia, nausea and fever. The last 2 are typical of post embolic syndrome common to all embolization procedures. The most frequent adverse events for surgery patients were dysuria and hematuria. Events also include non-TEAEs.
Time Frame: Through early termination of study (with less than 25% of subjects completing 12 month follow up)
Population: as for outcome 1
Measure: Number; unit: events per patient
Arm/Group | Prostate Artery Emoblization (PAE) | Transurethral Resection of the Prostate (TURP)
Number analyzed (Participants) | 28 | 6
events per patient
  Mild adverse events | 3.78 | 4.0
  Moderate adverse events | 0.39 | 0.5
  Severe adverse events | 0.21 | 0.17

5. Secondary Outcome: Number of Patients With Procedure Related Adverse Events
Description: Safety summaries will include the incidence of treatment-emergent adverse events (TEAEs). Treatment-emergent adverse events (TEAEs) are defined as any event that began on or after the date of treatment or worsened in severity or frequency after treatment was initiated. Events worsening in severity should be considered new adverse events. Adverse events recorded on the case report form (CRF) which began prior to treatment will not be included in the summary tables but will be included in the AE data listings.
Time Frame: TEAEs at time of study termination, with less than 25% of subjects completing 12 month follow up
Population: De Novo classification from FDA expanding the indication for Embosphere Microspheres to include prostatic artery embolization for symptomatic benign prostatic hyperplasia received 2017. IDE supplement proposed the termination of study follow-up visits; FDA granted approval of termination 03Nov2017. Early termination resulted in small numbers analyzed w less than 25% reaching 12 month follow-up.
Measure: Count of Participants; unit: Participants
Groups:
- Prostate Artery Embolization (PAE): Summary of treatment emergent adverse events presented as number of events in the PAE arm.
  Denominator for percent calculations is 52 treated subjects. Subjects who were randomized and never treated are not included.
  An AE is considered related to treatment if the Investigator assessment of relationship to study treatment was possible, probably, or definite.
  If a subject had multiple reports of the same type of AE, he is only counted once for that AE. System organ class counts are number of subjects.
- Transurethral Resection of Prostate (TURP): Summary of treatment emergent adverse events presented as number of events in the TURP arm.
  Denominator for percent calculations is 6 treated subjects. Subjects who were randomized and never treated are not included.
  An AE is considered related to treatment if the Investigator assessment of relationship to study treatment was possible, probably, or definite.
  If a subject had multiple reports of the same type of AE, he is only counted once for that AE. System organ class counts are number of subjects.
Arm/Group | Prostate Artery Embolization (PAE) | Transurethral Resection of Prostate (TURP)
Number analyzed (Participants) | 52 | 6
Participants
  Cardiac disorders | 3 | 1
  Congenital, familial and genetic disorders | 1 | 0
  Ear and labryinth disorders | 3 | 0
  Endocrine disorders | 1 | 0
  Gastrointestinal disorders | 22 | 2
  General disorders and administration site conditions | 11 | 0
  Infections and infestation | 7 | 1
  Injury, poisoning and procedural complications | 3 | 0
  Investigations | 1 | 1
  Metabolism and nutrition disorders | 2 | 0
  Musculoskeletal and connective tissue disorders | 10 | 1
  Nervous system disorders | 7 | 1
  Renal and urinary disorders | 30 | 5
  Reproductive system and breast disorders | 13 | 2
  Respiratory, thoracic and mediastinal disorders | 4 | 2
  Skin and subcutaneous tissue disorders | 3 | 2
  Surgical and medical procedures | 1 | 0
  Vascular disorders | 4 | 0

6. Other Pre Specified Outcome: Free Prostate Specific Antigen (PSA) at 6 Month Follow up
Description: Free PSA percentage summarized for both groups at 6 months follow up
Time Frame: 6 month follow up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Prostate Artery Emoblization (PAE) | Transurethral Resection of the Prostate (TURP)
Number analyzed (Participants) | 17 | 3
percentage | 18.7 (8.7) | 26.0 (8.7)

7. Other Pre Specified Outcome: Peak Urine Flow Rate (Qmax) at 1 Month
Description: The peak urine flow rate (Qmax) from the urodynamic and uroflowmetry assessments was assessed at 1 month follow up. (Additional timepoints were not assessed due to early termination).
Time Frame: 1 month follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL/s
Arm/Group | Prostate Artery Emoblization (PAE) | Transurethral Resection of the Prostate (TURP)
Number analyzed (Participants) | 23 | 4
mL/s | 12.1 (10.2) | 14.0 (4.1)

8. Other Pre Specified Outcome: International Index of Erectile Function (IIEF)
Description: Erectile Function (Questions 1-5 & 15), score range 0-5, max score = 30 Orgasmic Function (Questions 9-10), score range 0-5, max score = 10 Sexual Desire (Questions 11-12), score range 1-5, max score = 10 Intercourse Satisfaction (Questions 6-8), score range 0-5, max score = 15 Overall Satisfaction (Questions 13-14), score range 1-5, max score = 10
  SCORING for erectile dysfunction (Total of Q1-5 and Q15) is interpreted as follows:
  1-10: Severe Erectile Dysfunction 11-16: Moderate dysfunction 17-21: Mild to moderate dysfunction 22-25: Mild dysfunction 26-30: No dysfunction
  For all subscales, higher scores = less dysfunction/dissatisfaction Total IIEF is out of 75
Time Frame: 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Prostate Artery Emoblization (PAE) | Transurethral Resection of the Prostate (TURP)
Number analyzed (Participants) | 22 | 6
score on a scale
  Total IIEF (Q1 to 15 out of 75 points total) | 33.3 (24.4) | 61.7 (25.3)
  Erectile function (sub-score Q1-5, 15 out of total 30pts) | 12.6 (11.4) | 25.3 (11.4)
  Orgasmic function sub-score Q9-10 out of 10 points total) | 4.1 (4.0) | 7.3 (3.3)
  Sexual desire sub-score Q11-12 out of 10 points total | 5.9 (2.4) | 8.7 (2.4)
  Intercourse satisfaction sub-score Q6-8 out of 15 points total | 5.5 (5.8) | 11.7 (5.8)
  Overall satisfaction sub-score Q13-14 out of 10 points total | 5.4 (3.1) | 8.7 (3.3)

9. Other Pre Specified Outcome: Mean Prostate Volume, as Determined by MRI
Description: The mean prostate volume as assessed by MRI is summarized at 3 month time point.
Time Frame: 3 month follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Prostate Artery Emoblization (PAE) | Transurethral Resection of the Prostate (TURP)
Number analyzed (Participants) | 23 | 4
grams | 52.1 (15.0) | 28.2 (5.8)

10. Other Pre Specified Outcome: Post-void Residual Urinary Volume (PVR)
Description: The post void residual volume (PVR) from the urodynamic and uroflowmetry assessments is summarized for both treatment groups at 1 month time point.
Time Frame: 1 month follow-up
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Prostate Artery Emoblization (PAE) | Transurethral Resection of the Prostate (TURP)
Number analyzed (Participants) | 23 | 4
mL | 106 (136) | 7.5 (9.6)

11. Other Pre Specified Outcome: Total Prostate Specific Antigen (PSA) at 6 Months
Description: Prostate specific antigen (PSA) will be summarized for both treatment groups for 6 month time point
Time Frame: 6 months
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Prostate Artery Emoblization (PAE) | Transurethral Resection of the Prostate (TURP)
Number analyzed (Participants) | 19 | 4
ng/mL | 2.9 (2.0) | 2.1 (1.1)

ADVERSE EVENTS:
Time Frame: Study was intended to follow subjects through 12 months, but was terminated early due to de novo 510k clearance. Less than 25% of subjects reached the 12 month time point.
Description: Denominator for % calculations is 52 subjects in the PAE arm and 6 subjects in the TURP arm. Subjects randomized & never treated are not included.
  If a subject had multiple reports of same AE type, he is only counted once for that AE. System organ class counts = number of subjects.
Groups:
- Prostate Artery Embolization (PAE) Arm: Denominator for percent calculations is 52 treated subjects. Subjects who were randomized and never treated are not included. If a subject had multiple reports of the same type of AE, he is only counted once for that AE.
- Transurethral Resection of the Prostate (TURP) Arm: Denominator for percent calculations is 6 treated subjects. Subjects who were randomized and never treated are not included. If a subject had multiple reports of the same type of AE, he is only counted once for that AE.
Arm/Group | Prostate Artery Embolization (PAE) Arm | Transurethral Resection of the Prostate (TURP) Arm
All-Cause Mortality (participants affected / at risk) | 0/52 | 0/6
Serious Adverse Events (participants affected / at risk) | 6/52 | 1/6
Other Adverse Events (participants affected / at risk) | 40/52 | 5/6
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prostate Artery Embolization (PAE) Arm (N=52) | Transurethral Resection of the Prostate (TURP) Arm (N=6)
Impacted stool (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prostate Artery Embolization (PAE) Arm (N=52) | Transurethral Resection of the Prostate (TURP) Arm (N=6)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ear Pain (Ear and labyrinth disorders) | 3 (3) | 0 (0)
Catheter site inflammation (General disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Bladder injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Burning sensation (Nervous system disorders) | 1 (1) | 0 (0)
Bladder discomfort (Renal and urinary disorders) | 2 (2) | 0 (0)
Ejaculation disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Haematoma (Vascular disorders) | 1 (1) | 0 (0)
Bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Hypogonadism (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal rigidity (Gastrointestinal disorders) | 2 (2) | 0 (0)
Anorectal discomfort (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (3) | 1 (1)
Dental necrosis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 1 (1)
Haematochezia (Gastrointestinal disorders) | 3 (3) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 2 (2) | 1 (1)
Hiatal hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 8 (8) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)
Catheter site related reaction (General disorders) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Facial pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 0 (0)
Local swelling (General disorders) | 2 (2) | 0 (0)
Pain (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 3 (3) | 0 (0)
Suprapubic pain (General disorders) | 2 (2) | 0 (0)
Cellulits (Infections and infestations) | 1 (1) | 0 (0)
Localised infection (Infections and infestations) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (2)
Sepsis (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 4 (4) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Blood urine present (Investigations) | 1 (1) | 0 (0)
Urine leukocyte esterase positive (Investigations) | 0 (0) | 1 (1)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Chest wall mass (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (2) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 0 (0)
Presyncope (Nervous system disorders) | 2 (2) | 0 (0)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Sensory loss (Nervous system disorders) | 0 (0) | 1 (1)
Bladder spasm (Renal and urinary disorders) | 5 (5) | 0 (0)
Dysuria (Renal and urinary disorders) | 19 (23) | 3 (3)
Haematuria (Renal and urinary disorders) | 7 (7) | 3 (3)
Incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
Micturition (Renal and urinary disorders) | 4 (4) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0)
Terminal dribbling (Renal and urinary disorders) | 1 (1) | 0 (0)
Urethral pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 2 (2) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (2) | 0 (0)
Urinary straining (Renal and urinary disorders) | 1 (1) | 0 (0)
Epididymal cyst (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Haematospermia (Reproductive system and breast disorders) | 4 (4) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 5 (5) | 0 (0)
Penile burning sensation (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Penile pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Perineal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Prostatitis (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Retrograde ejaculation (Reproductive system and breast disorders) | 2 (2) | 1 (1)
Testicular pain (Reproductive system and breast disorders) | 1 (2) | 0 (0)
Varicocele (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin discoloration (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1)
Arthroscopic surgery (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Merit Medical received 513(f)(2) (de novo) classification from the FDA expanding the indication for Embosphere Microspheres to include prostatic artery embolization (PAE) for symptomatic benign prostatic hyperplasia (BPH) in 2017. An IDE supplement was submitted for this study proposing the termination of study follow-up visits. The FDA granted approval of termination on 03 Nov 2017. Early termination resulted in small numbers analyzed, incomplete enrollment and follow-up of study subjects.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-15): https://cdn.clinicaltrials.gov/large-docs/40/NCT01789840/Prot_SAP_000.pdf